CLINICAL TRIAL: NCT04391660
Title: Estimation of the Incidence of Colonization of Peripheral Venous Catheters After Skin Disinfection With 0.5% Sodium Hypochlorite, Preceded or Not by an Application of 70% Ethanol: Pilot, Monocentric, Randomized, Open-label Study
Brief Title: Estimation of the Incidence of Colonization of Peripheral Venous Catheters After Skin Disinfection With 0.5% Sodium Hypochlorite, Preceded or Not by an Application of 70% Ethanol
Acronym: DACLEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DACLEAN
Record Dates: First submitted 2020-05-06; First posted 2020-05-18 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-05

CONDITIONS: Skin Disinfection Before Peripheral Venous Catheter Insertion
MeSH Terms: interventions — Sodium Hypochlorite; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5% sodium hypochlorite solution (Active Comparator)
  Interventions: Drug: 0.5% sodium hypochlorite solution
- 0.5% sodium hypochlorite solution and 70% ethanol (Active Comparator)
  Interventions: Drug: 0.5% sodium hypochlorite solution and 70% ethanol

INTERVENTIONS:
Drug: 0.5% sodium hypochlorite solution — Disinfection with a 0.5% sodium hypochlorite solution applied with a sterile compress. This same antiseptic will be used at each dressing change.
  Arms: 0.5% sodium hypochlorite solution
Drug: 0.5% sodium hypochlorite solution and 70% ethanol — Disinfection with a 0.5% sodium hypochlorite solution applied with a sterile compress preceded by an application of 70% ethanol with a sterile compress, for its immediate bactericidal action. 0.5% sodium hypochlorite solution will be applied once the alcohol has evaporated and the skin is visually dried. These same antiseptics will be used at each dressing change.
  Arms: 0.5% sodium hypochlorite solution and 70% ethanol

SUMMARY:
The peripheral venous catheter is the most commonly used medical device in the hospital setting. Infectious complications are infrequent, bacterial or fungal, and local or systemic (catheter-related bacteremia). The latter prolong the length of hospitalization and increase the cost of care and mortality. For peripheral venous catheters, the risk of catheter-related bacteremia is lower (0.2-0.7 episodes per 1000 catheter days) than for other intravascular devices. However, the much higher number of peripheral venous catheters used explains a total number of infections close to that of other catheters. Colonization is usually the preliminary step to catheter infection. It is far more common than infection. Skin disinfection prior to catheter insertion is therefore essential to prevent this complication.

Currently, Chlorhexidine or Povidone Iodine in alcoholic solution is recommended before insertion of a peripheral venous catheter. Although rare, allergies may contraindicate these antiseptics. The widespread use of antiseptics in recent years for hand disinfection, mouthwashes or body baths could increase the risk of the development of strains that have become less sensitive, or even resistant, to currently available antiseptics. Allergies and reduced sensitivity require the search for alternatives to currently available solutions. Sodium hypochlorite is used to disinfect mucous membranes or healthy skin before an invasive procedure in children under 30 months of age. Very few studies have evaluated its efficacy in adults for this same indication, despite the fact that it was the first antiseptic used to prevent infections.

The aim of this study is to estimate the colonization rate of peripheral venous catheters after skin disinfection with 0.5% sodium hypochlorite (Dakin®) alone or preceded by an application of 70% ethanol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old) requiring hospitalization in participating services
* Having an indication for the placement of a peripheral venous catheter for an expected duration of at least 48 hours
* Free subject, without guardianship or curatorship or subordination
* A person affiliated to or benefiting from a social security scheme.
* Having given free and informed consent

Exclusion Criteria:

* Hypersensitivity to any of the constituents of Dakin® and/or Cooper® modified alcohol;
* History of epilepsy,
* Placement of a peripheral venous catheter in the emergency room that does not allow the usual rules of hygiene to be respected;
* Difficult vascular access foreseeable (drug addict, obese, non-visible veins...);
* Participation in another research protocol reducing the risk of catheter-related infection;
* Patient having received an antibiotic treatment in the 15 days prior to inclusion in the study;
* Patient who has already participated in the study;
* Subjects not affiliated with a Social Security system.
* Subjects benefiting from enhanced protection, namely persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection (guardianship and trusteeship) and finally patients in emergency situations.
* Pregnant or breastfeeding women, women of child-bearing age who do not have effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of colonized catheters | Up to 14 days

SECONDARY OUTCOMES:
Local infection, defined as colonization of the catheter or purulent discharge at the insertion site with a positive culture or no culture at the insertion site (a negative culture, in the absence of antibiotics, eliminates the case) | Up to 14 days
General infection, defined as colonization of the catheter in the presence of general signs of infection and total or partial regression of these signs within 48 hours after catheter removal | Up to 16 days
  General infection, defined as colonization of the catheter in the presence of general signs of infection (fever > 38.5° or hypothermia < 36°, chills, hypotension with PAS < 90 mmHg) and total or partial regression of these signs within 48 hours after catheter removal
Catheter-related bacteremia/fungemia | Up to 14 days
Incidence of a positive catheter culture regardless of the threshold and the microorganism under consideration | Up to 14 days
Incidence of local skin reaction and its severity | Up to 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Poitiers, Poitiers, France